CLINICAL TRIAL: NCT00208182
Title: Risperidone Monotherapy in the Treatment of PTSD in Women Survivors of Domestic Abuse and Rape Trauma: a Double-Blind, Placebo Controlled, Randomized Clinical Trial
Brief Title: Risperidone in the Treatment of PTSD in Women Survivors of Domestic Abuse and Rape Trauma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIS-USA-245B
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-03-10 (Estimated); Status verified 2006-03

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
This medical study is an assessment of clinical response in women with Posttraumatic Stress Disorder (PTSD) due to domestic violence or rape trauma when treated with risperidone. Response to risperidone or placebo (inactive drug) is measured by Clinician Administered PTSD Scale (CAPS) and Treatment Outcomes PTSD Scale (TOP-8). Second, the effect of risperidone on depressive and anxiety symptoms will be assessed using the Hamilton Rating Scale for Anxiety, Hamilton Rating Scale for Depression and the Clinical Global Impression.

DETAILED DESCRIPTION:
Risperidone is an atypical antipsychotic that has been shown to be effective in both the core PTSD symptoms and psychotic symptoms associated with combat-induced PTSD in males. Case series have shown that risperidone is possibly effective in monotherapy or adjunctively in treating PTSD patients. However, risperidone has never been tested in women with severe PTSD. Thus, we propose extending and expanding this research to another antipsychotic, risperidone, in a cohort of women who suffer PTSD as a consequence of domestic violence and/or rape trauma.

ELIGIBILITY:
Inclusion Criteria:

* Women with DSM-IV clinical diagnosis of PTSD caused by domestic violence or rape, who are able to attend weekly clinic appointments;
* Age 19 -64, not pregnant and either sterile or using acceptable contraception;
* A willingness and ability to provide competent signed informed consent;
* A level of understanding sufficient to perform all tests and examinations required by the protocol (including fluency of spoken English).

Exclusion Criteria:

* Any diagnosis of schizophrenia or bipolar I disorder; or active substance dependence.
* Unstable general medical condition or serious illness (e.g., death or hospitalization is anticipated within one year), poor liver or kidney function-Subjects with prior non-response to risperidone for the treatment of PTSD with an adequate trial
* Enrolment in any drug study within the last 60 days.
* Pregnancy or nursing.
* Any subject judged clinically to be at serious suicidal risk in the opinion of the investigator.

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2001-07; Study Completion 2004-08

PRIMARY OUTCOMES:
To compare the response in PTSD symptoms in women survivors of domestic violence or rape when treated with risperidone v. placebo, as measured by the Clinician Administered PTSD Scale (CAPS), and the TOP-8.

SECONDARY OUTCOMES:
To assess the effect of risperidone on depressive and anxiety symptoms in this study population. Instruments used include Hamilton Rating Scale for Anxiety, Hamilton Rating Scale for Depression and the Clinical Global Impression.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Petty, MD, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry and Research Center, Omaha, Nebraska, United States